CLINICAL TRIAL: NCT03116776
Title: Walnut Shell Glasses Moxibustion for Dry Eye Syndrome: a Randomized Controlled Trial
Brief Title: Walnut Shell Glasses Moxibustion for Dry Eye Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Weiwei Fu, Postgraduate, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-121-KY-01
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Dry Eye
Keywords: walnut shell glasses moxibustion; dry eye; randomized controlled trial
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: outcome assessor and statistician will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walnut Shell Glasses Moxibustion (Experimental): Use wire to make a glass frame which can fix two walnut shells and moxa roll in front of the eyes, the walnut shell should be soaked in medlar chrysanthemum water and use the moxibustion to treat eye disease.
  Interventions: Procedure: Walnut Shell Glasses Moxibustion
- Sodium hyaluronate eye drops (Active Comparator): Commonly used artificial tears in clinical.
  Interventions: Drug: Sodium hyaluronate eye drops

INTERVENTIONS:
Procedure: Walnut Shell Glasses Moxibustion — Participants in experimental group will receive 12 sessions of walnut shell glasses moxibustion, each for 30 minutes,3 times per week, and administered over 4 weeks.
  Arms: Walnut Shell Glasses Moxibustion
Drug: Sodium hyaluronate eye drops — One drop for each eye, four times per day for over 4 weeks.
  Arms: Sodium hyaluronate eye drops

SUMMARY:
This trial is designed to evaluate the efficacy of walnut shell glasses moxibustion for dry eye syndrome compared with sodium hyaluronate eye drops.

ELIGIBILITY:
Inclusion Criteria:

1. eyes are in line with dry eye diagnostic criteria.
2. Age 18 to 75 years,
3. signed informed consent, voluntary adherence to treatment for more than 1 month.

Exclusion Criteria:

1. combined with other eye disease (such as conjunctiva, cornea and iris have significant lesions).
2. eye surgery within 3 months.
3. pregnant or lactating women.
4. oral the drugs which could inhibit lacrimal gland secretion.
5. severe meibomian gland dysfunction.
6. severe eye burns, chemical injury patients.
7. combined with cardiovascular and cerebrovascular, liver, kidney and hematopoietic system and other serious primary disease, mental patients.
8. patients with Sjogren's syndrome.
9. patients who are participating in other drug clinical trials.
10. patients who are using other drugs or therapies for the treatment of dry eyes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
change from baseline in OSDI score | week 4, week 16, week 28
  We use the ocular surface disease index(OSDI) to evaluate the degree of dry eye. Assessing time point: at week 4, week 16, week 28.

SECONDARY OUTCOMES:
the efficacy of Walnut Shell Glasses Moxibustion | week 4, week 16, week 28
  The proportion of patients whose OSDI score reduced more than 50%
change from baseline in mean weekly OSDI score | week 1-4, week 16, week 28
  The mean weekly OSDI score over weeks 1-4 will be calculated as as the sum of each week divided by the number of weeks assessed.
change from baseline in VAS of eye discomfort | week 4, week 16, week 28
  Eye discomfort VAS scale: for the eye symptoms of self-assessment. Dry eye symptoms include itching, foreign body sensation, burning sensation, pain, dry, blurred vision, photophobia, eye swelling, tear Crack，ect. The overall discomfort are evaluate by VAS . Uses a 100-mm line that is labeled at each end. 0 mm represents no eye discomfort, 100 mm represents the most intolerable eye discomfort. Patient will rate the VAS(average VAS in the past 24h three times a week).
change from baseline in mean daily VAS score | week 1-4, week 16, week 28
  Patients will rate their average eye comfort with VAS three times a week. The mean daily VAS over week 1-4 will be calculated as the sum of each day divided by the number of days assessed.
change from baseline in BUT | week 2, week 4
  Check the tear break time(BUT) should be carried out before the other steps in the operation of the eye, used to evaluate the stability of the tear film. In the room without air flow, 1% of the sodium fluorescein with a glass rod dipped in a little coating in the lower eyelid conjunctival sac, the patient after several times, through the slit lamp cobalt blue light wide band inspection tear film, with a stopwatch Record the last time after the completion of the first blink of an eye to open to the tear film appeared in the first randomly distributed dry spots or black lines of time, recorded three times to take the mean.
change from baseline in SchimerⅠtext | week 2, week 4
  Evaluation the tear secretion, do not use ocular surface anesthetic, measuring the amount of reflex tear secretion. Place the test paper in the middle and outer 1/3 of the conjunctiva of the lower eyelid, and instruct the patient to lighten his eyes or look down at the bottom, and remove it after 5 minutes to measure the wetness from the beginning of the bend.
change from baseline in corneal fluorescence staining scores | week 2, week 4
  Corneal fluorescein staining: 2% fluorescein sodium coated with glass rods in the conjunctival sac, observed under the slit lamp to observe whether the corneal epithelium with staining, such as yellow-green stained, suggesting that corneal epithelial cell integrity damage. Score by 12 points. Cornea was divided into 4 quadrants, each quadrant was 0-3, no staining was 0, 1 to 30 dotted was 1 point, > 30 dotted but not fused For 2 points, 3 points for the emergence of corneal punctate staining, filaments and ulcers.
patiant's expectations for moxibustion | baseline
  This questionnaire includes three brief questions to investigate whether patients believe that moxibustion treatment will be useful. The relationship between patients' expectations and the effectiveness of moxibustion will be investigated because patients' beliefs about treatment enhanced or attenuated the effectiveness of treatment in a previous experimental study .

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei Fu, Principal Investigator — Department of Acupuncture, Guang' anmen hospital，China Academy of Chinese Medical Science, Beijing(100053), China
Locations (2):
- China (2):
  - Guang'anmen Hospital, China Academy of Chinese Medical Sceince, Beijing, Beijing Municipality
  - Guang'anmen Hospital, China Academy of Chinese Medical Science, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes